CLINICAL TRIAL: NCT04864821
Title: Clinical Study of CD276 Targeted Autologous Chimeric Antigen Receptor T Cell Infusion in Patients With CD276 Positive Advanced Solid Tumor
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA-P276-001
Record Dates: First submitted 2021-04-25; First posted 2021-04-29 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Osteosarcoma; Neuroblastoma; Gastric Cancer; Lung Cancer
MeSH Terms: conditions — Osteosarcoma; Neuroblastoma; Stomach Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- T cell injection targeting CD276 chimeric antigen receptor (Other)
  Interventions: Drug: Targeting CD276 CAR T cells

INTERVENTIONS:
Drug: Targeting CD276 CAR T cells — Targeting CD276 autologous chimeric antigen receptor T cells

SUMMARY:
Cd276 (B7-H3) is an ideal target for car-t treatment because of its high expression on the surface of neuroblastoma, osteosarcoma, gastric cancer and lung cancer cells, but not in normal peripheral cells or tissues. In conclusion, car-t cell therapy has achieved exciting results in blood tumors, but it has been stopped in solid tumor. The main reason for the poor effect is the existence of tumor microenvironment of solid tumor, which inhibits the chemotaxis and infiltration of car-t cells to tumor site. Therefore, in this clinical experiment, we will explore the best model of car-t therapy for solid tumor by intravenous and local tumor injection, which will bring new hope to patients with osteosarcoma, neuroblastoma and gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* The patients were aged from 1 to 70 years old (including the cut-off value), and the gender was not limited;
* The expected survival time was more than 12 weeks;
* ECoG score was 0-2;
* One of the following tumor types was confirmed by pathology: osteosarcoma, neuroblastoma, gastric cancer or lung cancer, and the positive rate of cd276 expression in tumor tissue was more than 50% by immunohistochemistry;
* Patients with ineffective standard treatment methods (such as postoperative recurrence, chemotherapy, radiotherapy, and progression after targeted drugs);
* According to RECIST 1.1, there was at least one measurable lesion (the longest diameter of solid lesion ≥ 10 mm, or the short diameter of lymph node lesion ≥ 15 mm);
* The function of main organs was normal (white blood cell count ≥ 3 × 109 / L, neutrophil count ≥ 1.5 × 109 / L, hemoglobin ≥ 8.5g/dl, platelet count ≥ 80 × 109 / L and lymphocyte count at 1 × 109 / L (including) ~ 4 × 109 / L (inclusive);
* The liver and kidney function and cardiopulmonary function meet the following requirements:

  1. Urea and serum creatinine ≤ 1.5 × ULN；
  2. Left ventricular ejection fraction ≥ 50%;
  3. Baseline oxygen saturation ≥ 94%;
  4. Total bilirubin ≤ 1.5 × ULN； ALT and AST ≤ 2.5 × ULN；
* The patient or legal representative can fully understand the significance and risk of this trial and has signed the informed consent.

Exclusion Criteria:

* Patients with history of immune deficiency or autoimmune diseases (including but not limited to rheumatoid arthritis, systemic lupus erythematosus, vasculitis, multiple sclerosis, insulin-dependent diabetes, etc.); Patients with graft-versus-host disease (GVHD) or need immunosuppressive agents;
* There was a history of other second malignancies in 5 years before screening;
* Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) were positive, and the peripheral blood HBV DNA titer was not within the normal reference value; HCV antibody and HCV RNA in peripheral blood were positive; HIV antibody positive patients; Syphilis was positive;
* Severe heart disease: including but not limited to unstable angina pectoris, myocardial infarction (within 6 months before screening), congestive heart failure (NYHA classification ≥ III), severe arrhythmia;
* Unstable systemic diseases judged by researchers: including but not limited to severe liver, kidney or metabolic diseases requiring drug treatment;
* Within 7 days before screening, there were active or uncontrollable infections requiring systemic treatment (except mild urogenital infection and upper respiratory tract infection);
* Pregnant or lactating women, female subjects who plan to conceive within one year after cell transfusion, or male subjects whose partners plan to conceive within one year after cell transfusion;
* Patients who had received car-t therapy or other gene modified cell therapy before screening;
* The subjects who were receiving systemic steroid treatment within 7 days before the screening or who needed long-term systemic steroid treatment (except inhalation or local use) were determined by the researchers;
* The ascites increased gradually after 2 weeks of conservative treatment (such as diuresis, sodium restriction, excluding ascites drainage);
* According to the judgment of the researcher, it does not conform to the situation of cell preparation;
* Other researchers think that it is not suitable for inclusion.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-14 (Estimated); Primary Completion 2022-05-14 (Estimated); Study Completion 2023-05-14 (Estimated)

PRIMARY OUTCOMES:
AE | 2 years after treatment
  adverse event
ORR | 12 weeks after treatment
  Objective remission rate
Cmax | 2 years after treatment
  The highest concentration of CAR-T cells in peripheral blood after infusion

IPD SHARING:
Plan to Share IPD: No